CLINICAL TRIAL: NCT01232686
Title: Snow Disease Surveillance System Study
Acronym: Snow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); The Royal Norwegian Ministry of Health (Other); Norwegian Health Network (state owned enterprise) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ID 3746/ HST954-10
Record Dates: First submitted 2010-10-15; First posted 2010-11-02 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2015-12

CONDITIONS: Communicable Diseases
Keywords: Communicable Diseases; Epidemiology; Population surveillance; Computerized Medical Record; Data collection
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control area (No Intervention): In the control areas we will monitor the prevalence and treatment of communicable diseases without giving the participants online access to disease surveillance information
- Intervention area (Experimental): In these areas we will give study participants online access to epidemiological data for communicable diseases
  Interventions: Other: Online disease surveillance data access

INTERVENTIONS:
Other: Online disease surveillance data access — In the intervention areas we will give the study participants online access to the Snow disease surveillance system. The system will provide data about the incidents of respiratory and gastrointestinal communicable diseases in the patient population.
  Arms: Intervention area

SUMMARY:
The study investigates whether shared online access to epidemiological data for general practitioners, disease prevention officers, emergency care services and microbiology laboratories changes clinical practice with regard to testing, diagnosing and treatment of communicable diseases. The main hypothesis is that "online access for general practitioner to epidemiological data about communicable diseases changes clinical practice for testing, diagnosing and treatment of communicable diseases".

DETAILED DESCRIPTION:
We will collect data from general practitioners (GP) offices by installing local data extraction solutions. Each installation will build a local anonymous database of GP consultations extracted from the local electronic patient record (EPR) system. These anonymous data records will be used to produce local disease statistics before they are exported to a centralized server available in the Norwegian Health network. The centralized server will produce daily reports about the epidemiological situation in the patient population. We will combine the syndromic data from the GP offices with data from the microbiology laboratories on the hospitals that covers the study areas. The epidemiological data will be made available to the intervention areas in the study through web based and customized client applications.

By using data extracted from the GP offices EPR databases and the microbiology laboratories we will investigate the study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering General Practitioner (GP) working in a GP office

Exclusion Criteria:

* The GP does not use a Electronic Patient Record (EPR) system

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Earlier diagnosis and treatment for communicable diseases | Measured at the end of the data collection period, approx. 1.5 year. (December 2012)
  General practitioners (GP) have three possible decisions in a consultation with a patient; 1) treat on suspicion, 2) take a sample, 3) wait and see whether the patient recovers or get worse, or 4) a combination of 1 and 2.
  In situations with decision 3 (wait and see) the patient may return to a consultation later on.
  The hypothesis is that online access to epidemiological data from the local patient population will enable GPs to make the right decision more often based on knowledge about the epidemiological situation in the patient population.

SECONDARY OUTCOMES:
Earlier detection of local disease outbreaks | Measured at the end of the data collection period, approx. 1.5 year. (December 2012)
  Syndromic surveillance enables earlier detection of local disease outbreaks compared to traditional laboratory based surveillance. We will record the time of disease outbreak detection in both intervention and control areas and compare.
Lower number of infected during disease outbreaks | Measured at the end of the data collection period, approx. 1.5 year. (December 2012)
  We will compare the number of infected in the intervention and control areas. The hypothesis is that the intervention areas will have fewer infected compared to the control areas.
Impact on health service costs | Measured at the end of the data collection period, approx. 1.5 year. (December 2012)
  We will measure the cost related to communicable diseases in the control and intervention areas. Our prediction is that it will change.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Gustav Bellika, PhD, Principal Investigator — University of Tromsø, Department of Computer Science